CLINICAL TRIAL: NCT05218447
Title: Dosing of Overground Robotic Gait Training with Functional Outcomes and Neuroplasticity After Spinal Cord Injury
Acronym: DOOR SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Texas Woman's University (Unknown)
Responsible Party: Principal Investigator, Chad Swank, Research Investigator, Baylor Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BSWRI IRB 021-205
Record Dates: First submitted 2021-12-20; First posted 2022-02-01 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-09

CONDITIONS: Spinal Cord Injuries
Keywords: Exoskeleton; Wearable assistive technology; Transcranial magnetic stimulation; Robotic gait training
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned into one of 4 gait training groups: usual care (UC) gait training only; high frequency RGT - 4 sessions/week for 6 weeks; moderate frequency RGT - 3 sessions/week for 8 weeks; or low frequency RGT - 2 sessions/week for 12 weeks
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: All clinical and study specific assessments will be completed by trained assessors blinded to group allocation. Clinical assessments will be completed by a physical therapist (e.g., WISCI-II, SCIM). Study specific assessments (e.g., FSS, actigraphy, TMS) will be conducted by study staff and investigator. Subjects will not be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Low Frequency (Experimental): Subjects will receive 2 sessions of robotic gait training (RGT) per week for 12 weeks
  Interventions: Device: Robotic Gait Training
- Moderate Frequency (Experimental): Subjects will receive 3 sessions of robotic gait training (RGT) per week for 8 weeks
  Interventions: Device: Robotic Gait Training
- High Frequency (Experimental): Subjects will receive 4 sessions of robotic gait training (RGT) per week for 6 weeks
  Interventions: Device: Robotic Gait Training
- Control Group (Active Comparator): Subjects will receive usual care gait training without robotic gait training
  Interventions: Other: Usual Care (UC) Gait Training

INTERVENTIONS:
Device: Robotic Gait Training — Subjects will be randomized to one of 4 gait training group. The duration of treatment will span across their inpatient rehabilitation length of stay after providing informed consent to their 9 months post-SCI visit in the outpatient rehabilitation setting.
  Subjects will wear an exoskeleton device and receive robotic gait training (RGT) with a physical therapist during a 45-minutes inpatient rehabilitation session. Subjects will complete 24 robotic gait training sessions over different durations during outpatient rehabilitation. Subjects will also complete a transcranial magnetic stimulation (TMS) assessment and questionnaires about walking and function. Subjects will be asked to wear an activity monitor to measure their activity.
  Other Names: Ekso GT™ robotic exoskeleton
  Arms: High Frequency; Low Frequency; Moderate Frequency
Other: Usual Care (UC) Gait Training — Subjects will be randomized to one of 4 gait training group. The duration of treatment will span across their inpatient rehabilitation length of stay after providing informed consent to their 9 months post-SCI visit in the outpatient rehabilitation setting.
  Subjects will complete gait training with a physical therapist during a 45-minutes inpatient rehabilitation session. Subjects will also complete a transcranial magnetic stimulation (TMS) assessment and questionnaires about walking and function. Subjects will be asked to wear an activity monitor to measure their activity.
  Arms: Control Group

SUMMARY:
The DOOR SCI project examines dosing effects of robotic gait training (RGT) and transcranial magnetic stimulation (TMS) initiated during inpatient rehabilitation and continued through early outpatient rehabilitation

DETAILED DESCRIPTION:
Emerging evidence indicates that robotic exoskeleton use results in positive outcomes for those with chronic SCI, yet limited evidence exists for the acute setting. The potential benefit of RGT initiated during inpatient rehabilitation when recovery is greatest is unknown yet appears promising due to established principles of neuroplasticity and the fact that RGT incorporates the critical components of gait training. As a result of the lack of evidence, no clinical practice guidelines exist that delineate which gait retraining approach or dose during early phases of recovery results in the best outcomes for people with motor incomplete SCI. The DOOR SCI project examines dosing effects on 5 occasions over 9 months: (1) inpatient rehabilitation admission and (2) discharge, (3) after completing 24 RGT sessions, (4) 1-month post RGT, and (5) 9-months post SCI). To test the overarching goal, investigators propose three specific aims:

Aim 1: Using a randomized controlled trial, prospectively examine whether the dosing frequency [24 sessions delivered as high, moderate, or low frequency, defined by number days/week (4, 3, or 2 days/week over 6, 8, 12 weeks)] of RGT therapy provided during the acute/subacute recovery phase after motor incomplete SCI impacts outcomes compared to usual care only.

Aim 2: Investigate the difference over 9 months of the neuroplastic effect of RGT dosing as measured by single pulse TMS.

Aim 3: Evaluate the safety, tolerability, and feasibility of delivering different dosing frequencies of RGT from inpatient to outpatient rehabilitation settings.

ELIGIBILITY:
Inclusion Criteria:

* All types of motor incomplete SCI (traumatic and non-traumatic)
* Acute/Subacute phase of recovery
* Medically stable as deemed by physician
* Undergoing medical care and rehabilitation at Baylor Scott & White Institute for Rehabilitation
* Both genders and all races and ethnicities
* Meet the Ekso robotic exoskeleton frame limitations
* Continence of or a program for bladder and bowel management

Exclusion Criteria:

* Concurrent moderate to severe traumatic brain injury (TBI)
* Degenerative diagnoses
* Pre-morbid developmental disability, significant psychological diagnosis, or other cognitive impairment
* Pregnancy

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2025-06-14 (Estimated); Study Completion 2025-09-14 (Estimated)

PRIMARY OUTCOMES:
Change in Walking Index for Spinal Cord Injury - II (WISCI-II) from baseline | Change in baseline, within 5 days of discharge, within 5 days post-intervention (RGT Groups) or 1-month post-discharge (UC group), 1-month post-intervention or 2-months post-discharge (UC group) (5) 9-months post-SCI onset
  The WISCI-II defines the physical limitation for gait secondary to impairment at the person level and indicates the ability of a person to walk after SCI. The WISC-II rank orders the ability a person to walk on a scale of 0-20 with 0 representing no ability to stand or participate in assisted walking and 20 representing an ability to walk 10 meters with no devices, no braces, and no physical assistance.

SECONDARY OUTCOMES:
Change in 10-Meter Walk Test (10MWT) | Change in baseline, within 5 days of discharge, within 5 days post-intervention (RGT Groups) or 1-month post-discharge (UC group), 1-month post-intervention or 2-months post-discharge (UC group) (5) 9-months post-SCI onset
  The 10MWT assesses gait speed (m/s) over a short duration.
Change in Spinal Cord Independence Measure (SCIM) | Change in baseline, within 5 days of discharge, within 5 days post-intervention (RGT Groups) or 1-month post-discharge (UC group), 1-month post-intervention or 2-months post-discharge (UC group) (5) 9-months post-SCI onset
  The SCIM assesses the ability of a person with spinal cord injury (SCI) to preform specified tasks independently, with assistance, or with assistive devices.
  SCIM is composed of 19 items with total SCIM scores ranging from 0 (required assistance) to 100 (independence). A higher score means greater independence.
Change in Numerical Pain Rating Scale (NPRS) | Change in baseline, within 5 days of discharge, within 5 days post-intervention (RGT Groups) or 1-month post-discharge (UC group), 1-month post-intervention or 2-months post-discharge (UC group) (5) 9-months post-SCI onset
  Pain is a significant problem in many individuals with SCI. A 0-10 Point Numerical Pain Rating Scale (NRS) is recommended as the outcome measure for pain intensity after SCI during acute and subacute phases. Pain severity can be categorized into 3 distinct groups as relates to pain interference: 1-3 (mild), 4-7 (moderate), 8-10 (severe). A higher score means greater pain severity.
Change in Fatigue Severity Scale (FSS) | Change in baseline, within 5 days of discharge, within 5 days post-intervention (RGT Groups) or 1-month post-discharge (UC group), 1-month post-intervention or 2-months post-discharge (UC group) (5) 9-months post-SCI onset
  The Fatigue Severity Scale (FSS) is used to measure fatigue in neurologic disorders and measures the effects of fatigue on function. It is measure on the following scale:
  1. - Strongly Disagree
  2. - Disagree
  3. - Slightly Disagree
  4. - Neutral
  5. - Slightly Agree
  6. - Agree
  7. - Strongly Agree A higher score means greater fatigue.
Change in Penn Spasm Frequency Scale (PSFS) | Change in baseline, within 5 days of discharge, within 5 days post-intervention (RGT Groups) or 1-month post-discharge (UC group), 1-month post-intervention or 2-months post-discharge (UC group) (5) 9-months post-SCI onset
  The PSFS is a self-report measure to assess a patient's perception of spasticity frequency and severity following a SCI. With excellent internal consistency (ICC = 0.90), the current version was modified from the original to include both frequency and severity. A higher score means greater magnitude in spasms.
Change in Patient Health Questionnaire - 9 (PHQ-9) | Change in baseline, within 5 days of discharge, within 5 days post-intervention (RGT Groups) or 1-month post-discharge (UC group), 1-month post-intervention or 2-months post-discharge (UC group) (5) 9-months post-SCI onset
  The PHQ-9 is a self-report measure to assess the presence of depressive symptoms. Each items is scored on the following scale:
  0 - not at all
  1. - several days
  2. - more than half the days
  3. - nearly daily
  Total scores are calculated by adding all the score and provides a possible depression severity score:
  none (0-4), mild (5-9), moderate (10-14), moderately severe (15-19), and severe (20-27). A higher score means greater severity in depressive symptoms.
Change in Life Satisfaction Questionnaire (LISAT) | Change in baseline, within 5 days of discharge, within 5 days post-intervention (RGT Groups) or 1-month post-discharge (UC group), 1-month post-intervention or 2-months post-discharge (UC group) (5) 9-months post-SCI onset
  The LISAT is a nine-item quality of life questionnaire suitable for SCI populations containing a single item assessing overall life satisfaction, along with eight additional domain-specific items. Items are answered on a 6-point likert scale that ranges from 1 (very dissatisfied), to 6 (very satisfied). The total Life Satisfaction score is computed as the mean of the item scores and the results are divided into dissatisfied (1-4) and satisfied (5-6). A higher score score means greater life satisfaction.
Change in Physical Activity by GT9x Actigraph accelerometer | Change in baseline, within 5 days of discharge, within 5 days post-intervention (RGT Groups) or 1-month post-discharge (UC group), 1-month post-intervention or 2-months post-discharge (UC group) (5) 9-months post-SCI onset
  Active energy expenditure will be measured in counts per day using a GT9x Actigraph accelerometer. Patient will be instructed to wear the watch on an unaffected wrist for one week. Higher counts represent greater physical activity.
Change in Neurophysiologic biomarkers by single pulse transcranial magnetic stimulation (TMS) | Change in baseline, within 5 days of discharge, within 5 days post-intervention (RGT Groups) or 1-month post-discharge (UC group), 1-month post-intervention or 2-months post-discharge (UC group) (5) 9-months post-SCI onset
  Motor evoked potential (MEP) amplitudes will be measured and indexed from lower extremity muscle by single pulse transcranial magnetic stimulation (TMS).

OTHER OUTCOMES:
Rate of adverse events | Through study completion, an average of 9 months
  Number of adverse events occurring at baseline through study completion.
Self-reported tolerance of treatment | Through study completion, an average of 9 months
  Subjects provide feedback on their tolerance of treatment sessions via an 18-item questionnaire. The questionnaire measures tolerability on a scale 0 (Not tolerable at all to 10 (Maximally tolerable). A higher score means greater tolerability in robotic gait training.
Rate of treatment completion | Through study completion, an average of 9 months
  The average number of session attended divided by the number of scheduled sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Swank, PhD, PT, NCS, Principal Investigator — Baylor Research Institute
Locations (1):
- Baylor Scott & White Institute for Rehabilitation, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swank C, Trammell M, Bennett M, Ochoa C, Callender L, Sikka S, Driver S. The utilization of an overground robotic exoskeleton for gait training during inpatient rehabilitation-single-center retrospective findings. Int J Rehabil Res. 2020 Sep;43(3):206-213. doi: 10.1097/MRR.0000000000000409. PMID 32282573
- [Background] Swank C, Sikka S, Driver S, Bennett M, Callender L. Feasibility of integrating robotic exoskeleton gait training in inpatient rehabilitation. Disabil Rehabil Assist Technol. 2020 May;15(4):409-417. doi: 10.1080/17483107.2019.1587014. Epub 2019 Mar 19. PMID 30887864
- [Background] DiPasquale J, Trammell M, Clark K, Fowler H, Callender L, Bennett M, Swank C. Intensity of usual care physical therapy during inpatient rehabilitation for people with neurologic diagnoses. PM R. 2022 Jan;14(1):46-57. doi: 10.1002/pmrj.12577. Epub 2021 Apr 15. PMID 33599119
- [Background] Swank C, Galvan C, DiPasquale J, Callender L, Sikka S, & Driver D. Lessons Learned with Robotic Exoskeleton Use During Rehabilitation - therapeutic and medical severity considerations. Technology & Disability. 2020; 32(2): 103-110.
- [Derived] Suhalka A, da Silva Areas FZ, Meza F, Ochoa C, Driver S, Sikka S, Hamilton R, Goh HT, Callender L, Bennett M, Shih HT, Swank C. Dosing overground robotic gait training after spinal cord injury: a randomized clinical trial protocol. Trials. 2024 Oct 18;25(1):690. doi: 10.1186/s13063-024-08503-0. PMID 39425122